CLINICAL TRIAL: NCT00219024
Title: An 8 Week Double-blind, Multicenter, Randomized, Multifactorial, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of Aliskiren Administered Alone and in Combination With Hydrochlorothiazide in Patients With Essential Hypertension
Brief Title: Clinical Study to Evaluate the Efficacy and Safety of Aliskiren Alone and in Combination With Hydrochlorothiazide in Patients With Essential Hypertension.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2204
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Hypertension
Keywords: Hypertension, aliskiren, blood pressure, hydrochlorothiazide (HCTZ).
MeSH Terms: conditions — Hypertension | interventions — aliskiren

INTERVENTIONS:
Drug: aliskiren

SUMMARY:
To demonstrate the efficacy and safety of aliskiren given to patients with essential hypertension, at doses of 75 mg, 150 mg and 300 mg alone, and in combination with hydrochlorothiazide (HCTZ)

ELIGIBILITY:
Inclusion Criteria

* Patients with essential hypertension
* Patients who are eligible and able to participate in the study

Exclusion Criteria

* Severe hypertension
* History or evidence of a secondary form of hypertension
* History of hypertensive encephalopathy or cerebrovascular accident

Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2775 (Actual)
Dates: Start 2004-08; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in diastolic blood pressure after 8 weeks

SECONDARY OUTCOMES:
Change from baseline in systolic blood pressure after 8 weeks
Diastolic blood pressure is < 90 mmHg or a reduction from baseline of > 10 mmHg after 8 weeks
Blood pressure < 140/90 mmHg
Change from baseline in standing diastolic blood pressure after 8 weeks
Change from baseline in standing systolic blood pressure after 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States
- Investigative Centers, Germany

REFERENCES:
- [Derived] Yan JH, Jarugula V, Sabo R, Papst CC, Zhang J, Dole WP. Pharmacokinetics and pharmacodynamics of aliskiren/hydrochlorothiazide single-pill combination tablets and free combination of aliskiren and hydrochlorothiazide. J Clin Pharmacol. 2012 May;52(5):645-55. doi: 10.1177/0091270011405499. Epub 2011 Jun 9. PMID 21659626